CLINICAL TRIAL: NCT06908083
Title: A Study to Evaluate Immunologic and Virologic Parameters During Analytical Treatment Interruption Following Combination bNAb Therapy During Suppressive ART
Brief Title: Immunologic and Virologic Parameters During Analytical Treatment Interruption Following Combination bNAb Therapy During Suppressive ART
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10002295; 002295-I
Record Dates: First submitted 2025-04-01; First posted 2025-04-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01-15

CONDITIONS: HIV
Keywords: HIV Infection; Analytical Treatment Interruption; bnab therapy
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults living with HIV (Experimental): Participants who received either two intravenous infusions of 3BNC117-LS (dosed at 30 mg /kg) and 10-1074-LS (dosed at 10 mg/kg) or two saline infusions (placebo) at weeks 0, and 20 as part of the Rockefeller University trial (MCA-1034) or the NIH trial (001037) and are willing to interrupt treatment and then restart once criteria is met.
  Interventions: Other: Analytical Treatment Interruption

INTERVENTIONS:
Other: Analytical Treatment Interruption — Participants will stop their ART (Antiretroviral therapy) on Week 0 and will remain off of their ART for up to 48 weeks or until they meet restart criteria.

SUMMARY:
Background:

Recent studies have shown bNAbs may help remove cells that are infected with HIV (HIV reservoir) from the body and may also change how the immune system fights HIV.

Objective:

The purpose of this research study is to see if and when HIV levels in the blood (viral load) rise after the participant stops their HIV medication. We will also measure the highest number (peak) of the virus before each participant starts their HIV medications again. For most people treated with standard HIV medications, the HIV virus amount will increase within 2 to 4 weeks after stopping their HIV medications. This study is only open to participants who have taken part in an earlier study (MCA-1034 or NIH number 001037). In the earlier study, participants either received a combination of 3BN117-LS and 10-1074-LS (two anti-HIV monoclonal antibodies) OR received placebo (salt water). In this new study, researchers will compare the participants who received the antibodies to those who did not to see what effect the antibodies may have had on the HIV reservoir.

Researchers will also look at:

* side effects people may have when they stop their HIV medications.
* changes in the number of blood cells carrying inactive HIV (the HIV reservoir size).
* the blood cells that can clear HIV before, following temporarily stopping, and after re-starting HIV medications.
* how well HIV may be controlled after a participant stops their HIV medication.

Eligibility:

People aged 18 to 70 years with HIV who completed protocol MCA-1034 (NIH Study 001037).

Design:

Participants will be screened. They will have a physical exam. They will answer questions about their health. Blood samples will be taken.

Participants will stop their HIV medications for a period of time. They will have blood tests every 2 weeks and clinic visits every 4 weeks for 24 weeks to check their HIV levels and to make sure they are not having side effects. There will be strict safety rules for restarting HIV medications. Some participants whose HIV levels remain low at 24 weeks may continue without ART for another 24 weeks; they will have blood tests every 2 to 4 weeks.

Participants may undergo leukapheresis up to 3 times: Leukapheresis is a several hours long procedure in which blood is collected from a vein in one arm, processed through an attached machine, and then returned to the person through a vein in the opposite arm.

Participants will have 4 follow-up visits over 24 weeks after they restart ART.

Participants will remain in the study up to 18 months.

DETAILED DESCRIPTION:
Study Description:

This is an exploratory study to evaluate virologic and immunologic parameters during analytical treatment interruption (ATI) in people

with HIV (PWH) who participated in protocol MCA-1034 (NIH # 001037), which evaluated HIV-1 reservoir dynamics in peripheral blood during combination bNAb therapy plus ART or ART alone. MCA-1034 participants will be invited to participate in this study after completing all MCA-1034 follow up visits. MCA-1034 treatment assignment will not be known at enrollment in this study until unblinding of MCA-1034 occurs. Under MCA-1034, participants will have received two intravenous infusions of 3BNC117-LS (dosed at 30 mg/kg) and 10-1074-LS (dosed at 10 mg/kg) or placebo at weeks 0 and 20 while on standard ART and will have completed 80 weeks of follow up after the first antibody infusions. Participants will be eligible to enter this study from 12 to 24 weeks after the last MCA-1034 study visit.

Participants who enroll in this study will discontinue ART at study entry (week 0/day 0) and will be followed every other week until meeting pre-defined ART restart criteria. The ATI period will last up to 24 weeks (Step 1 weeks 0-24). Participants who do not meet ART restart criteria will be offered to remain off ART until meeting ART restart criteria for up to 24 additional weeks with monitoring every 4 weeks, unless HIV-1 RNA is >= 200 copies/ml when monitoring will occur every 2 weeks (Step 2 weeks 25-48; i.e. maximum ATI period of 48 weeks).

At the end of the ATI period, all participants will be advised to resume ART even if they have not experienced return of viremia. Participants who experience return of viremia and/or meet ART resumption criteria will be followed for 24 weeks after resuming ART.

Objectives:

Primary Objectives:

- To evaluate the kinetics of plasma viral rebound during ATI in PWH who participated in protocol MCA-1034 (NIH # 001037) and received combination bNAb or placebo during suppressive ART.

Secondary Objectives:

* To evaluate the occurrence of adverse events following ART discontinuation.
* To evaluate changes in HIV-1 reservoir size in peripheral blood prior to, following ATI and after re-initiation of ART.
* To evaluate HIV-1 specific cellular immune responses prior to, following ATI and after re-initiation of ART.
* To evaluate levels of immune exhaustion and immune activation prior to, following ATI and after re-initiation of ART.

Exploratory Objectives:

* To evaluate the degree (magnitude) of plasma viral rebound during ATI in PWH who participated in protocol MCA-1034 (NIH # 001037) and received combination bNAb or placebo during suppressive ART.
* To characterize the HIV-1 reservoir clonal composition in peripheral blood prior to, following ATI and after re-initiation of ART.
* To characterize host HIV-1 specific humoral and cellular immune responses prior to, following ATI and after reinitiation of ART.
* To genotypically and phenotypically characterize plasma rebound viruses.
* To correlate virologic outcomes with bNAb sensitivity of reservoir proviruses.
* To correlate virologic and immunologic outcomes with time to meeting ART restart criteria.

Endpoints: Primary Endpoint:

- The difference in the time to meet criteria to restart ART between protocol MCA-1034 bNAb and placebo recipients.

Secondary Endpoints:

* The difference in peak plasma viremia from ART discontinuation to meeting ART restart criteria between protocol MCA-1034 bNAb and placebo recipients.
* The occurrence of grade 3 or higher adverse events (AE) (including confirmed laboratory abnormalities) that are possibly, probably, or definitely related to ART discontinuation.
* The occurrence of serious adverse events, regardless of relationship to ART discontinuation.
* Change in the intact proviral reservoir size, measured by droplet digital PCR (ddPCR) or intact proviral deoxyribonucleic acid assay (IPDA) prior to, following ATI and after re-initiation of ART.
* Changes in HIV-1 specific T cell immune responses in peripheral blood, measured by enzyme-linked immunospot (ELISpot) or intracellular cytokine staining (ICS) prior to, following ATI and after re-initiation of ART.
* Changes in immune exhaustion and immune activation cellular or soluble markers by flow cytometry or by ELISA methods prior to, following ATI and after re-initiation of ART.

Exploratory Endpoints:

* Clonal composition of the intact proviral reservoir before and after immunotherapy with 3BNC117-LS and 10-1074-LS during suppressive ART by quadruplex polymerase chain reaction (Q4PCR) or other appropriate assays that may become available prior to, following ATI and after re-initiation of ART.
* HIV-1 transcriptional activity as determined by spliced and unspliced HIV-1 ribonucleic acid (RNA) in circulating total CD4+ T cells and/or other appropriate assays prior to, following ATI and after re-initiation of ART.
* Changes in HIV-1 specific T cell immune responses in peripheral blood, measured by assays such as epitope mapping, proliferation and viral inhibition assays prior to, following ATI and after re-initiation of ART.
* Changes in binding capacity and neutralizing activity of autologous antibody responses to pre-ATI and post-ATI proviruses and rebound plasma viruses.
* Env sequencing and neutralization sensitivity of plasma rebound viruses to 3BNC117-LS, 10-1074-LS and autologous IgG by TZM/bl.
* Correlation between bNAb sensitivity of baseline proviruses (i.e. MCA-1034 entry) and virological outcomes (e.g. time to meeting ART restart criteria and peak viremia during ATI).
* Correlation between pre-ATI virological (e.g. proviral reservoir size and transcriptional activity) and immunological measures (e.g. magnitude, breadth and functionality of HIV-1 specific T cell immune responses, and autologous neutralization titers) and time to meeting ART restart criteria.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability to provide informed consent;
2. Stated willingness to comply with all study procedures and availability for the duration of the study;
3. Adult persons of any sex, aged 18 years to 70;
4. Participated in Protocol MCA-1034 (NIH # 001037) and completed follow up 12 to 24 weeks prior to study entry (day 0);
5. On antiretroviral therapy with plasma HIV-1 RNA levels of less than or equal to 50 copies/ml and no reported interruption of ART for 7 consecutive days or longer for at least 48 weeks.

   NOTE: A single plasma HIV-1 RNA >50 copies/mL but less than 200 copies/mL that is followed by an HIV-1 RNA <= 50 copies/mL is permitted;
6. Current CD4+ T cell counts >= 400 cells/mcL, CD4+ T cell % >= 15%;
7. If on an NNRTI-based regimen, willing to switch to an integrase or protease inhibitor-based regimen for at least 4 weeks prior to discontinuing ART;
8. For participants who can become pregnant (i.e., participants who have not been post-menopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy), negative pregnancy test at screening and within 48 hours prior to entry.

   NOTE: Participant-reported history is acceptable as documentation of hysterectomy and bilateral oophorectomy, tubal ligation, tubal micro-inserts, and vasectomy;
9. Participants who can become pregnant must agree to use one method of contraception, from the highly effective methods for contraception listed below. Barrier methods of contraception are permitted as a method of contraception. Contraception must be used from study entry and until ART is reinitiated and viral suppression is achieved. Acceptable methods of contraception include:

   * Condom with spermicide
   * Diaphragm with spermicide
   * Contraceptive subdermal implant
   * Intrauterine device or intrauterine system
   * Combined estrogen and progestogen oral contraceptive
   * Injectable progestogen
   * Contraceptive vaginal ring
   * Percutaneous contraceptive patches Partner sterilization with documentation of azoospermia prior to the participant's entry into the study, and this partner is the sole partner for that participant, will be allowed. The documentation of partner sterility can come from the site personnel's review of medical records, medical examination and/or semen analysis, or medical history interview provided by the participant or the partner. Self-reported documentation of reproductive potential should be entered in the source documents;
10. Willingness to use barrier protection (male or female) during sexual activity during ATI and until viral re-suppression for those who re-start ART.

EXCLUSION CRITERIA:

Any individual who meets any of the following criteria will be excluded from participation in this study:

1. History of AIDS-defining illness and/or known CD4 nadir less than 100 cells/mcL in the last 3 years;
2. History of systemic corticosteroids (e.g. an equivalent dose of prednisone of >20 mg daily for >14 days), immunosuppressive anti-cancer, interleukins, systemic interferons, systemic chemotherapy or other medications considered significant by the trial physician within the last 3 months;
3. Any clinically significant acute or chronic medical condition (e.g. such as autoimmune diseases, cirrhosis, active malignancy that may require systemic chemotherapy or radiation therapy), other than HIV infection, that in the opinion of the investigator would preclude participation;
4. History of or current clinical atherosclerotic cardiovascular disease (ASCVD), as defined by 2018 ACC/AHA guidelines, including a previous diagnosis of any of the following:

   * Acute myocardial infarction
   * Acute coronary syndromes
   * Stable or unstable angina
   * Coronary or other arterial revascularization procedures
   * Stroke
   * Transient ischemic attack
   * Peripheral arterial disease presumed to be of atherosclerotic origin;
5. Any history of an HIV-associated malignancy, including Kaposi's sarcoma, or any type of lymphoma or virus-associated cancers;
6. Any history of Progressive Multifocal Leukoencephalopathy (PML);
7. Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the preceding 36 months or for whom such therapies are expected in the subsequent 12 months; NOTE: minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) is not exclusionary.
8. Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or isolated positive HBV core antibody or hepatitis C virus RNA (HCV-RNA) in blood; NOTE: Participants with a positive test for HCV antibody and a negative test for HCV RNA are eligible; as are participants with isolated HBcAb who are receiving an ART regimen that do not include tenofovir (TAF or TDF).
9. Pregnancy or lactation;
10. Receipt of cabotegravir-LA IM or rilpivirine-LA IM within 24 months prior to study entry.
11. Documented multiclass antiretroviral drug resistance that, in the judgment of the investigator, would pose a risk of virologic failure should additional mutations develop during the study;
12. Laboratory abnormalities in the parameters listed below:

    * Absolute neutrophil count <1,000 cells/mcl;
    * Hemoglobin <10 gm/dL;
    * Platelet count <100,000 cells/mcl;
    * ALT >1.5 x ULN;
    * AST >1.5 x ULN;
    * Total bilirubin greater than 1.5 x ULN;
    * eGFR <60 mL/min/1.73m^2;
13. Receipt of an investigational product within 12 weeks prior to study entry or expected participation in such a study during this study.
14. Participation in other studies that require frequent blood sample collection during participation in this study.
15. Active drug or alcohol use or any other pattern of behavior that, in the opinion of the investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to Restart ART | Week 0 until Week 48 or when participant meets restart criteria
  Difference in number of days from stopping ART (Day 0) until participant meets restart criteria between MCA-1034/001037 (NIH) bNAb and placebo recipients

SECONDARY OUTCOMES:
Difference in Peak Plasma Viremia | Week 0 until Week 48 or when participant meets restart criteria
  Number of grade 3 or higher adverse events that occur during Analytical Treatment The difference in peak plasma viremia from Week 0 until week 48 or when participant meets restart criteria between MCA-1034/001037 (NIH) bNAb and placebo recipients
Frequency of Grade 3 or higher Adverse Events | Week 0 until Week 48 or when participant meets restart criteria
  Number of grade 3 or higher adverse events that occur during Analytical Treatment Interruption that are possibly, probably, or definitely related.
Frequency of Serious Adverse Events | Week 0 until Week 48 or when participant meets restart criteria
  Number of serious adverse events that occur during the Analytical Treatment Interruption regardless of relatedness
Change in intact proviral reservoir size | Throughout
  Change in the intact proviral reservoir size, measured by droplet digital PCR (ddPCR) or intact proviral deoxyribonucleic acid assay (IPDA) prior to, following ATI, and after re-initiation of ART.
Changes in HIV-1 Specific T Cell Immune Responses in Peripheral Blood | Throughout
  Changes in HIV-1 specific T cell immune responses in peripheral blood, measured by enzyme-linked immunospot (ELISpot) or intracellular cytokine staining (ICS) prior to, following ATI, and after re-initiation of ART.
Changes in immune exhaustion and immune activation cellular or soluble markers | Throughout
  Changes in immune exhaustion and immune activation cellular or soluble markers by flow cytometry or by ELISA methods prior to, following ATI, and after re-initiation of ART.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Rockefeller Institute, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be deposited at ImmPort. All laboratory findings will include unique, anonymized patient-level identifiers, patient age category, and HIV status/disease details including stage of disease, plasma viremia, and CD4 counts. High-quality sequencing data will be deposited into the Gene Expression Omnibus repository. Lower coverage sequences will be deposited into Zenodo or another general-purpose open data repository. Sanger and next-generation genomic and virus sequencing data will be deposited in GenBank or BioProject repository. Per informed consent documents in each protocol, de-identified raw data may be shared internally for research purposes as deemed appropriate by the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within one year of primary completion date of final subject

REFERENCES:
- [Background] Clarridge KE, Blazkova J, Einkauf K, Petrone M, Refsland EW, Justement JS, Shi V, Huiting ED, Seamon CA, Lee GQ, Yu XG, Moir S, Sneller MC, Lichterfeld M, Chun TW. Effect of analytical treatment interruption and reinitiation of antiretroviral therapy on HIV reservoirs and immunologic parameters in infected individuals. PLoS Pathog. 2018 Jan 11;14(1):e1006792. doi: 10.1371/journal.ppat.1006792. eCollection 2018 Jan. PMID 29324842
- [Background] Sneller MC, Huiting ED, Clarridge KE, Seamon C, Blazkova J, Justement JS, Shi V, Whitehead EJ, Schneck RF, Proschan M, Moir S, Fauci AS, Chun TW. Kinetics of Plasma HIV Rebound in the Era of Modern Antiretroviral Therapy. J Infect Dis. 2020 Oct 13;222(10):1655-1659. doi: 10.1093/infdis/jiaa270. PMID 32443148
- [Background] Sneller MC, Blazkova J, Justement JS, Shi V, Kennedy BD, Gittens K, Tolstenko J, McCormack G, Whitehead EJ, Schneck RF, Proschan MA, Benko E, Kovacs C, Oguz C, Seaman MS, Caskey M, Nussenzweig MC, Fauci AS, Moir S, Chun TW. Combination anti-HIV antibodies provide sustained virological suppression. Nature. 2022 Jun;606(7913):375-381. doi: 10.1038/s41586-022-04797-9. Epub 2022 Jun 1. PMID 35650437
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002295-I.html